CLINICAL TRIAL: NCT01181154
Title: Rituximab in Adult's Warm Auto-Immune Hemolytic Anemia : a Phase III, Double-bind, Randomised Placebo-controlled Trial
Brief Title: Rituximab in Auto-Immune Hemolytic Anemia
Acronym: RAHIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P080704; 2008-008255-42 (EudraCT Number)
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Warm Autoimmune Hemolytic Anemia
Keywords: Auto-Immune; Hemolytic; Anemia; AHA; AIHA; Rituximab
MeSH Terms: conditions — Hemolysis; Anemia | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- equivalent volume total (=1000 ml) (Placebo Comparator): Placebo : equivalent volume total (=1000 ml)
  Interventions: Drug: Placebo
- rituximab (Mabthera®) (Experimental): rituximab (Mabthera®), 1000 mg at day 1 and day 15
  Interventions: Drug: rituximab (Mabthera®)

INTERVENTIONS:
Drug: rituximab (Mabthera®) — 1000 mg at day 1 and day 15
  Other Names: rituximab (Mabthera®)1000 mg at day 1 and day 15
  Arms: rituximab (Mabthera®)
Drug: Placebo — equivalent volume total
  Other Names: Placebo equivalent volume total
  Arms: equivalent volume total (=1000 ml)

SUMMARY:
The hypothesis based on retrospective data is that, the rate of overall response-rate (PR + CR) at 1 year will be much higher in the rituximab arm (80%) than in the placebo arm (20%).Thirty four patients (17 in each arm) will be include (amendment n°6 - 15/10/2013) over a 3 year period (amendment n°3 - 11/12/2012).

DETAILED DESCRIPTION:
The primary aim of the study is to assess the efficacy (overall response rate at 1 year) of rituximab (an anti-CD20 monoclonal antibody) in AIHA due to warm autoantibody when administered at the initial phase of the disease. All eligible patents with a newly diagnosed AIHA (within 6 weeks after diagnosis) will be treated by corticosteroids at standard dose (prednisone 1 mg/kg/day) and will be randomized into 2 arms: Rituximab or placebo 1000 mg on days 1 and 15 in a 1/1 ratio. As soon as at least a partial remission (PR) of AIHA will be achieved, the daily dose of prednisone will be tapered following the rules provided by the protocol.

The hypothesis based on retrospective data is that, the rate of overall response-rate (PR + CR) at 1 year will be much higher in the rituximab arm (80%) than in the placebo arm (20%).Thirty four patients (17 in each arm) will be include (amendment n°6 - 15/10/2013) over a 3 year period (amendment n°3 - 11/12/2012).

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. AIHA defined at time of diagnosis by a Hgb level £ 10 g/dL, with a reticulocytes count > 120 109/L, signs of hemolysis (at least a haptoglobin level < 4 mg/L), and a positive direct antiglobulin test (DAT) ( IgG or IgG + complement pattern).
3. Disease duration equal or less than 6 weeks at time of inclusion --> removed by amendment n°4 and substituted by :First episode of AIHA to "hot" antibody previously untreated or treated corticosteroids for less than 6 weeks.
4. Patients with an associated autoimmune thrombocytopenia (Evans' syndrome) will be eligible for the study if the platelet count is over 30 x 109/L at inclusion.
5. Normal level gammaglobulins in the serum (i.e. >5g/L) at inclusion.
6. Absence of detectable lymph nodes on a total body CT-scan (to be performed before inclusion if not performed at diagnosis).
7. Effective means of contraception during treatment and for six months after completion of treatment for all women of child bearing age
8. Negative serum pregnancy test within 14 days prior to study entry.
9. Written informed consent

Exclusion Criteria:

Previous treatment with rituximab

1. AIHA diagnosed and treated more than 6 weeks prior to inclusion removed by amendment n°4 and substituted by AIHA relapsed or newly diagnosed but treated with corticosteroids for more than 6 weeks
2. Ongoing immunosuppressive therapy (other than corticosteroids) or previous treatment administered within 2 weeks prior to the beginning of the study treatment
3. Non-Hodgkin Lymphoma (NHL) other than stage A chronic lymphoid leukemia
4. Previous or concomitant malignancy other than basal cell or squamous cell carcinoma of the skin, carcinoma-in-situ of the cervix, or other malignancy for which the patient had not been disease-free for at least 5 years.
5. Autoimmune disorder such as SLE with at least one extra-hematological manifestation requiring a treatment with steroids and/or immunosuppressive drugs.
6. Any other associated cause congenital or acquired hemolytic anemia (except thalassemia trait or heterozygous sickle cell anemia).
7. Negative DAT or DAT positive with isolated anti-C3d pattern related to the presence of a monoclonal IgM with cold agglutinin properties.
8. Positive HIV test and/or hepatitis virus C infection and/or positive hepatitis B virus surface antigen (HbsAg).
9. Neutrophils count < 1,000/mm 3 at inclusion.
10. Impaired renal function as indicated by a serum creatinine level > 2 mg/d
11. Inadequate liver function as indicated by a total bilirubin level > 2.0 mg/dL and/or an AST or ALT level > 2x upper limit of normal.
12. New York Heart Classification III or IV heart disease.
13. Previous history of severe psychiatric disorder or are unable to comply with study and follow-up procedures
14. Pregnant or lactating women, or woman planning to become pregnant within 12 months of receiving study drug
15. Absence of written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-03-03 (Actual); Primary Completion 2015-01-08 (Actual); Study Completion 2016-01-08 (Actual)

PRIMARY OUTCOMES:
Overall response rate (complete and partial response) in both arms | at 1 year

SECONDARY OUTCOMES:
Comparison in both arms of the mean cumulative doses of prednisone | at 1 year
Comparison in both arms of the number of transfusions of packed red blood cells in both arms | at 1 year
Comparison in both arms of the number of days in hospital | within the first year of follow-up
Comparison in both arms of the number of patients requiring a splenectomy and/or an immunosuppressor | during the first 12 months of follow-up
Comparison in both arm of the mortality | at 1 year
Comparison in both arm of overall response (CR + PR) | at 2 years
Comparison of the incidence of serious side effects in both arms | at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marc MICHEL, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor University Hospital, Créteil, France